CLINICAL TRIAL: NCT03887247
Title: Reducing Concurrent Opioid-Benzodiazepine Prescriptions Through Provider Intervention
Brief Title: Reducing Concurrent Opioid-Benzodiazepine Prescriptions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: United States Department of Defense (U.S. Federal Agency); General Services Administration (GSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REDUCE-CONCURRENT
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Adverse Drug Effect of Opioids; Adverse Drug Effect of Benzodiazepines
Keywords: Care coordination; Opioid; Benzodiazepine; Behavioral science; Behavioral economics; Nudge; Fragmentation of care; Concurrent prescribing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- E-Mail Alert (Active Comparator): Send email to the patient's opioid prescriber(s), benzodiazepine prescriber(s), and/or primary care manager.
  Interventions: Behavioral: E-mail Alert
- As-Usual (No Intervention): As-usual (no email) approach.

INTERVENTIONS:
Behavioral: E-mail Alert — Encrypted email to the following providers: the patient's opioid prescriber(s), benzodiazepine prescriber(s), and/or primary care manager. If there is more than one provider, they are copied together on the same message. The email identifies the concurrent prescriptions, details the patient's prescription history, includes relevant VA/DoD guidelines, states the risk of concurrent prescribing to patient, and provides action steps and relevant resources. When multiple providers are involved, the message encourages the providers to coordinate with each other and provides provider contact information to facilitate this communication.
  Arms: E-Mail Alert

SUMMARY:
The purpose of this effort is to use informative e-mails to improve the process of prescribing of opioids and benzodiazepines within the National Capital Region/Military Health System (NCR/MHS), with the aim of decreasing concurrent opioid and benzodiazepine prescribing.

DETAILED DESCRIPTION:
The purpose of this effort is to use low-cost informative e-mails to improve the process of prescribing of opioids and benzodiazepines within the National Capital Region/Military Health System (NCR/MHS), with the aim of decreasing concurrent opioid and benzodiazepine prescribing. Both the VA/DoD Clinical Practice Guideline for Opioid Therapy for Chronic Pain (2017) and the CDC Guideline for Prescribing Opioids for Chronic Pain (2016) strongly recommend against the concurrent use of opioids and benzodiazepines. Taken together, these drugs could cause respiratory depression, enhanced sedation, and death. The intervention population will be prescribers and primary care managers associated with patients who have recently received concurrent prescriptions of opioids and benzodiazepines. Using a randomized approach, we will allocate the NCR/MHS providers associated with patients with concurrent prescriptions for opioids and benzodiazepines to one of two conditions:

1. E-mail alert - A messaging approach, in which we will send encrypted emails to the patient's opioid and benzodiazepine prescriber(s) and primary care manager that identify the concurrent prescriptions and detail the patient's prescription history, inform them of the VA/DoD guideline and risk to patient, and provide action steps and relevant resources. When multiple providers are involved, the email message will also encourage coordination across providers and provide relevant contact information
2. As-Usual - An as-usual approach, in which providers are not sent messages. These providers can access patient information through the MHS Opioid Registry as before.

ELIGIBILITY:
Inclusion Criteria:

* Patient had an overlapping opioid-benzodiazepine prescription
* At least one of the patient's providers (opioid prescribers, benzodiazepine prescribers, and/or PCM) is in the NCR

Exclusion Criteria:

* Patient has a cancer diagnosis
* Patient is receiving palliative care
* Patient is under 18
* Patient was previously allocated to a study condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2234 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2021-07-29 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Overlapping Days | 90 days
  Overlapping days of opioids and benzodiazepines, determined using the dates of service and days supply of the prescription drug fills
Opioid Days | 90 days
  Days of opioids received
Benzodiazepine Days | 90 days
  Days of benzodiazepines received

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Brutcher, PharmD,PhD, Principal Investigator — Walter Reed National Military Medical Center and Uniformed Services University of the Health Sciences; Alan Sim, PhD, Principal Investigator — Defense Health Agency; Elana Safran, MPP, Principal Investigator — General Services Administration (GSA); Adam Sacarny, PhD, Principal Investigator — General Services Administration and Columbia University; Mary Steffel, PhD, Principal Investigator — General Services Administration and Northeastern University; Christopher J Spevak, MD, MPH, JD, Principal Investigator — Walter Reed National Medical Medical Center
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sacarny A, Safran E, Steffel M, Dunham JR, Abili OD, Mohajeri L, Oh PT, Sim A, Brutcher RE, Spevak C. Effect of Pharmacist Email Alerts on Concurrent Prescribing of Opioids and Benzodiazepines by Prescribers and Primary Care Managers: A Randomized Clinical Trial. JAMA Health Forum. 2022 Sep 2;3(9):e223378. doi: 10.1001/jamahealthforum.2022.3378. PMID 36218952